CLINICAL TRIAL: NCT02412254
Title: Aging, Cognition, and Hearing Evaluation in Elders Pilot Study
Brief Title: Aging, Cognition, and Hearing Evaluation in Elders Study
Acronym: ACHIEVE-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00067383; R34AG046548 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hearing intervention (Active Comparator): Best practices hearing rehabilitative treatment
  Interventions: Other: Best practices hearing rehabilitative treatment
- Successful aging intervention (Placebo Comparator): Successful aging intervention
  Interventions: Other: Successful aging intervention

INTERVENTIONS:
Other: Best practices hearing rehabilitative treatment — Intervention comprises hearing needs assessment, counselling, sensory management with amplification devices, and rehabilitative training.
  Arms: Hearing intervention
Other: Successful aging intervention — One-on-one education sessions on healthy aging topics (cancer screening, smoking cessation, etc.) between a trainer and participant
  Arms: Successful aging intervention

SUMMARY:
The investigators will conduct a small pilot study that will randomize ~ 40 70-84 year-old adults with hearing loss to best-practices hearing rehabilitative treatment (hearing assessment, counseling, fitting of amplification devices) versus a successful aging intervention (one-on-one counseling/education sessions on successful aging topics). Participants will be followed for 6 months, and outcomes will focus on communication, quality of life, cognition, and other functional surveys. This pilot study is in preparation for a larger planned trial to investigate if hearing loss treatment can reduce cognitive decline and dementia in older adults.

ELIGIBILITY:
Inclusion Criteria

* Age 70-84 years.
* Community-dwelling.
* Fluent English-speaker.
* Residency. Participants must plan to reside in the local area for the study duration (6 months).
* Audiometric hearing impairment. Participants must have adult-onset hearing impairment with a pure tone average (0.5, 1, and 2 kHz) in the better-hearing ear of ≥ 30 decibels and <70 dB.
* Word Recognition in Quiet score >60% bilaterally.
* Mini-Mental State Exam (MMSE) score ≥ 23 for individuals with high-school degree or less; Mini-Mental State Exam (MMSE) score ≥ 25 for individuals with some college or more
* Willingness to participate. Participants must be willing and able to consent to participate in the study, be willing to be randomized to either the Hearing intervention or to the Successful Aging intervention, and be willing to follow the study protocol for the duration of the trial.

Exclusion Criteria

Potential candidates for enrollment who meet one or more of t he following criteria are excluded from participation in the study:

* Self-reported disability in ≥ 2 or more Activities of Daily Living (ADL)
* Self-reported hearing aid use in the past year (>5 hours/week).
* Vision impairment (worse than 20/40 on MN Near Vision Card).
* Medical contraindication to use of hearing aids (e.g., draining ear).
* Conductive hearing impairment as determined by a difference in air audiometry and bone audiometry ("air-bone gap") greater than 15 dB in 2 or more contiguous frequencies in both ears.
* Unwilling to wear hearing aids on a regular (i.e., daily or near daily) basis
* No participants are excluded based on race or sex

Ages: 70 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE) | 6 month follow-up

SECONDARY OUTCOMES:
Neurocognitive test battery including Trail Making Test, Delayed Word Recall, and other tests | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lin, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Comstock Center for Public Health Research, Hagerstown, Maryland, United States

REFERENCES:
- [Derived] Deal JA, Albert MS, Arnold M, Bangdiwala SI, Chisolm T, Davis S, Eddins A, Glynn NW, Goman AM, Minotti M, Mosley T, Rebok GW, Reed N, Rodgers E, Sanchez V, Sharrett AR, Coresh J, Lin FR. A randomized feasibility pilot trial of hearing treatment for reducing cognitive decline: Results from the Aging and Cognitive Health Evaluation in Elders Pilot Study. Alzheimers Dement (N Y). 2017 Jun 21;3(3):410-415. doi: 10.1016/j.trci.2017.06.003. eCollection 2017 Sep. PMID 29067347